CLINICAL TRIAL: NCT04515784
Title: Examination of a Safety Aid Reduction Protocol for Treatment Resistant PTSD Among Veterans
Brief Title: Safety Aid Reduction Treatment for PTSD Among Veterans
Acronym: START-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHBP-003-19F
Record Dates: First submitted 2020-08-03; First posted 2020-08-17 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Safety aid; Treatment; Posttraumatic Stress Disorder; Veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: One-arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): Active arm- START-PTSD
  Interventions: Behavioral: Safety Aid Reduction Treatment for PTSD

INTERVENTIONS:
Behavioral: Safety Aid Reduction Treatment for PTSD — START-PTSD includes many of the key elements found in empirically supported treatments for PTSD including: a) psychoeducation regarding the development and maintenance of PTSD; and b) exposure to internal sensations and external situations that are connected to one's fear/distress response via identification and elimination of safety aids. Known safety aids to be covered include: cognitive avoidance (e.g., using mental distractions to avoid trauma-related images); situational avoidance (e.g., avoiding crowded market places); checking behaviors (e.g., checking doors, windows, locks, and perimeters more often than necessary); reassurance seeking (e.g., excessively watching the news); other compulsive behaviors (e.g., checking the location of exits); use of companions (e.g., relying on someone to attend a social gathering); and use of alcohol and certain substances (e.g., consuming alcohol to reduce anxiety).

SUMMARY:
The purpose of this project is to examine the acceptability, feasibility, and utility of a safety aid reduction treatment (START) among Veterans with posttraumatic stress disorder (PTSD). It is hypothesized that START will be acceptable, feasible, and will lead to reductions in PTSD symptom severity immediately and over time.

DETAILED DESCRIPTION:
Rates of posttraumatic stress disorder (PTSD) among military personnel have surged in recent years. In response, the Department of Veterans Affairs (VA) has launched nationwide training initiatives to disseminate two PTSD treatments with strong empirical support: prolonged exposure (PE) therapy and cognitive processing therapy (CPT). Despite the well-documented effectiveness of PE and CPT, only a minority of Veterans with PTSD initiate these trauma-focused treatments. One approach to addressing PTSD in a non-trauma-focused fashion is to utilize empirically supported treatments focused on safety aid reduction. Safety aids are maladaptive cognitive and/or behavioral strategies designed to prevent, avoid, or alleviate anxiety. Initially introduced as a way to explain how pathological anxiety can persist despite repeated exposure to feared stimuli, safety aids have been found to play a critical role in the etiology and maintenance of various anxiety and related conditions including PTSD. Importantly, a separate line of research suggests that safety aids are amenable to change through cognitive behavioral interventions. Although promising, these trials did not include patients with PTSD. In this context, the purpose of this project is to examine the acceptability, feasibility, and utility of a safety aid reduction treatment (START) for PTSD. Participants will include veterans with a diagnosis of PTSD who decline to participate in evidence-based psychotherapies (EBPs) for PTSD, namely PE or CPT. It is hypothesized that START will be acceptable, feasible, and will lead to reductions in PTSD symptom severity immediately and over time.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care at New Orleans VA
* Veterans with diagnosis of PTSD who decline trauma focused treatment

Exclusion Criteria:

* Substance dependence requiring detoxification
* Active psychosis
* Uncontrolled Bipolar Disorder
* Severe suicidal intent requiring hospitalization
* Current engagement in psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in PTSD diagnostic status as measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline and one-month follow-up
  The CAPS-5 is a 30-item clinician-administered interview designed to assess current (i.e., past month) and lifetime PTSD diagnostic status. In addition to assessing the 20 DSM-5 PTSD symptoms, the CAPS-5 contains questions regarding the onset and duration of symptoms, associated impairment in various life domains, and specifications for the dissociative subtype. The past month CAPS-5 will be administered at baseline and one-month follow-up to assess changes in PTSD diagnostic status.
Change in PTSD symptoms as measured by the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline, post-intervention (10-weeks), and one-month follow-up
  The PCL-5 is a 20-item self-report questionnaire designed to assess each of the 20 DSM-5 PTSD symptoms. Veterans will be asked to read a list of symptoms and indicate their level of distress as it relates to each within the past month using a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (Extremely) with higher scores reflecting increased symptom severity. The PCL-5 will be administered at baseline, immediately following the 10-week group, and at a one-month follow-up to assess changes in PTSD symptom severity.
Changes in safety aid usage as measured by the Safety Behavior Assessment Form (SBAF) | Baseline, post-intervention (10-weeks), and one-month follow-up
  The SBAF is a 41-item self-report questionnaire designed to assess safety behavior usage. Veterans will be asked to read a list of behaviors and rate how often they engage in each behavior using a 4-point Likert-type scale ranging from 0 (Never) to 3 (Always) with higher scores reflecting increased symptom severity. The SBAF will be administered at baseline, immediately following the 10-week group, and at a one-month follow-up to assess changes in safety behavior usage.
Client Satisfaction Questionnaire-8 (CSQ-8) | Post-intervention (10-weeks)
  The CSQ-8 is an 8-item self-report questionnaire designed to assess overall satisfaction with treatment services. Although response options differ from item-to-item, all questions are rated on a 4-point Likert-type scale ranging from 1 to 4 with higher scores indicating higher treatment satisfaction. The CSQ-8 will be administered immediately following the 10-week group to assess treatment acceptability.

SECONDARY OUTCOMES:
Changes in anxiety as measured by the Beck Anxiety Inventory (BAI) | Baseline, post-intervention (10-weeks), and one-month follow-up
  The BAI is a 21-item self-report questionnaire designed to assess the experience of anxiety symptoms. Veterans will be asked to rate how often they experience each symptom using a 4-point Likert-type scale ranging from 0 (Not at all) to 3 (Severely) with higher scores reflecting increased symptom severity. The BAI will be administered at baseline, immediately following the 10-week group, and at a one-month follow-up to assess changes in anxiety symptoms.
Changes in depression as measured by the Beck Depression Inventory-II (BDI-II) | Baseline, post-intervention (10-weeks), and one-month follow-up
  The BDI-II is a 21-item self-report questionnaire designed to assess symptoms associated with depression. Using a 4-point Likert-type scale ranging from 0 to 3, Veterans will be asked to select the statement from a group of statements that best represents how they have felt over the last two weeks with higher scores reflecting increased symptom severity. The BDI-II will be administered at baseline, immediately following the 10-week group, and at a one-month follow-up to assess changes in depression symptoms.
Changes in PTSD cognitions as measured by the Posttraumatic Cognitions Inventory (PTCI) | Baseline, post-intervention (10-weeks), and one-month follow-up
  The PTCI is a 33-item self-report questionnaire designed to assess trauma-related thoughts and beliefs including negative cognitions regarding the self, others, and the world. Veterans will be asked to read a list of statements and indicate the degree to which they agree or disagree with each statement using a 7-point Likert-type scale ranging from 1(totally disagree) to 7 (totally agree) with higher scores reflecting increased symptom severity. The PTCI will be administered at baseline, immediately following the 10-week group, and at a one-month follow-up to assess changes in PTSD cognitions.
Changes in funtional impairment as measured by the Sheehan Disability Scale (SDS) | Baseline, post-intervention (10-weeks), and one-month follow-up
  The SDS is a 3-item self-report questionnaire designed to assess functional impairment functional impairment in work/school, social, and family life. For each domain, Veterans will be asked to provide an impairment rating ranging from 0 (Not at all) to 10 (Extremely) with higher scores reflecting increased impairment. The SDS will be administered at baseline, immediately following the 10-week group, and at a one-month follow-up to assess changes in functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Raines, PhD, Principal Investigator — Southeast Louisiana Veterans Health Care System, New Orleans, LA
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to disclose data outside of the VA, however, if there is a need to disclose data outside of the VA (e.g., a member of the scientific community requests a copy), IRB approval will be sought, data will be de-identified prior to disclosing, and the disclosure will be recorded on a VA disclosure log as required by VA policy.

REFERENCES:
- [Background] Rosen CS, Bernardy NC, Chard KM, Clothier B, Cook JM, Crowley J, Eftekhari A, Kehle-Forbes SM, Mohr DC, Noorbaloochi S, Orazem RJ, Ruzek JI, Schnurr PP, Smith BN, Sayer NA. Which patients initiate cognitive processing therapy and prolonged exposure in department of veterans affairs PTSD clinics? J Anxiety Disord. 2019 Mar;62:53-60. doi: 10.1016/j.janxdis.2018.11.003. Epub 2018 Nov 20. PMID 30550959
- [Background] Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clin Psychol Rev. 2010 Aug;30(6):635-41. doi: 10.1016/j.cpr.2010.04.007. Epub 2010 May 2. PMID 20546985
- [Background] Dunmore E, Clark DM, Ehlers A. Cognitive factors involved in the onset and maintenance of posttraumatic stress disorder (PTSD) after physical or sexual assault. Behav Res Ther. 1999 Sep;37(9):809-29. doi: 10.1016/s0005-7967(98)00181-8. PMID 10458046
- [Background] Riccardi CJ, Korte KJ, Schmidt NB. False Safety Behavior Elimination Therapy: A randomized study of a brief individual transdiagnostic treatment for anxiety disorders. J Anxiety Disord. 2017 Mar;46:35-45. doi: 10.1016/j.janxdis.2016.06.003. Epub 2016 Jun 18. PMID 27397584
- [Background] Schmidt NB, Buckner JD, Pusser A, Woolaway-Bickel K, Preston JL, Norr A. Randomized controlled trial of false safety behavior elimination therapy: a unified cognitive behavioral treatment for anxiety psychopathology. Behav Ther. 2012 Sep;43(3):518-32. doi: 10.1016/j.beth.2012.02.004. Epub 2012 Mar 9. PMID 22697441
- [Background] Monson CM, Schnurr PP, Resick PA, Friedman MJ, Young-Xu Y, Stevens SP. Cognitive processing therapy for veterans with military-related posttraumatic stress disorder. J Consult Clin Psychol. 2006 Oct;74(5):898-907. doi: 10.1037/0022-006X.74.5.898. PMID 17032094
- [Background] Fulton JJ, Calhoun PS, Wagner HR, Schry AR, Hair LP, Feeling N, Elbogen E, Beckham JC. The prevalence of posttraumatic stress disorder in Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans: a meta-analysis. J Anxiety Disord. 2015 Apr;31:98-107. doi: 10.1016/j.janxdis.2015.02.003. Epub 2015 Feb 19. PMID 25768399

DOCUMENTS (1):
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT04515784/ICF_000.pdf